CLINICAL TRIAL: NCT03343483
Title: The Getting Active Project (GAP): A Randomized Trial of Volunteering to Reduce Loneliness in Later Life
Brief Title: The Helping Older People Engage Project: Improving Social Well-Being in Later Life
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kimberly Van Orden, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AG054457 (NIH); R01AG054457 (NIH)
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Loneliness; Quality of Life
Keywords: Volunteerism; Aged; Loneliness; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volunteering (Experimental): Structured social volunteering program providing peer companionship to frail, homebound older adults for at least 16 hours per month for 12 months.
  Interventions: Behavioral: Volunteering
- Life Review (Active Comparator): Self-guided program of life review for 12 months.
  Interventions: Behavioral: Life Review

INTERVENTIONS:
Behavioral: Volunteering — Volunteers provide non-medical caregiving for frail seniors-"care receivers"-to help them maintain their independence and improve their well-being. Friendly visiting is the primary service provided. Structured, intensive training is provided prior to placement. The target expectation is of interactions in person and/or by telephone for at least 16 hours per month. On-going training ("booster sessions") as well as volunteer support groups, and educational activities are provided. Participants not interested in serving as peer companions are allowed other volunteer options as long as the activities are deemed 'social' by the volunteer coordinator and are options routinely provided as part of the AmeriCorps Senior RSVP Program. COVID update: due to physical distancing requirements, volunteer placements have transitioned to remote friendly calling/letter writing or activities that can be conducted with physical distancing, such as delivery for Meals on Wheels.
  Arms: Volunteering
Behavioral: Life Review — Subjects will complete a self-guided life review exercise over 12 months. Subjects will complete one section of the life review (with the self-help book) each month and send 'assignments' once per month to an email 'counselor' who will respond with supportive comments within three days.
  Arms: Life Review

SUMMARY:
Older adults who feel lonely carry increased risk for reduced quality of life, morbidity, and mortality. Volunteering is a promising intervention for reducing loneliness in later life. The primary objective of this proposal is to test the hypothesis that a social volunteering program for lonely older adults will lead to reduced loneliness and improved quality of life.

This study compares the effect of a Senior Corps volunteering intervention versus a self-guided life review active control condition on feelings of loneliness in older adults.

The study involves randomly assigning older adults (150 women, 150 men) who report loneliness to 12 months of either: 1) a structured social volunteering program, or 2) an active control intervention with self-guided life review. Specific aims are as follows: 1) To examine the effect of volunteering on loneliness and quality of life; 2) To examine social engagement, perceived usefulness, and social support as mechanisms for reducing loneliness; 3) To examine conditions under which volunteering is most effective at reducing loneliness.

DETAILED DESCRIPTION:
The many negative outcomes associated with loneliness in older people have rendered loneliness itself a new public health target. Older adults who feel lonely carry increased risk for reduced quality of life, morbidity, and mortality. The risk of premature mortality related to loneliness is at least as large as the risks arising from such factors as obesity, physical inactivity, alcohol misuse, and smoking. Volunteering is a promising intervention for reducing loneliness in later life. The primary objective of this proposal is to test the hypothesis that a social volunteering program for lonely older adults will lead to reduced loneliness and improved quality of life. National infrastructure for volunteering (The Senior Corps) ensures that volunteering is a highly scalable intervention.

The investigators propose to compare the effect of a Senior Corps volunteering intervention versus a self-guided life review active control condition on feelings of loneliness in older adults. The investigators' preliminary data, as well as published studies of volunteering in later life, strongly suggest that volunteering should reduce loneliness. Rigorous experimental study is needed, however, to examine volunteering in both men and women who are lonely, to determine conditions that maximize benefit, and to understand mechanisms. The investigators hypothesize, per tenets of Self-Determination Theory, that increased social engagement and feelings of both usefulness and social support function as psychological mechanisms whereby volunteering reduces loneliness. Understanding these mechanisms will promote effective implementation, allowing communities to adapt volunteering programs while retaining the active ingredients.

The study involves randomly assigning older adults (150 women, 150 men) who report loneliness to 12 months of either: 1) a structured social volunteering program, or 2) an active control intervention with self-guided life review.

Specific aims are as follows: 1) To examine the effect of volunteering on loneliness and quality of life; 2) To examine social engagement, perceived usefulness, and social support as mechanisms for reducing loneliness; 3) To examine conditions under which volunteering is most effective at reducing loneliness.

The volunteering intervention is already implemented nation-wide, indicating high feasibility of going to scale (http://www.nationalservice.gov/programs/senior-corps). If effective, volunteering should be "prescribed" by physicians and promoted by policy. Dissemination and scaling up efforts will involve connecting primary care patients and aging services clients who are lonely with The Senior Corps, shown to be feasible in the investigators' companion study, The Senior Connection. Existing infrastructure will make it possible to reach a large proportion of lonely older adults. Reducing loneliness has the potential to improve well-being and save lives.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* English-speaking
* UCLA Short Form Loneliness Scale score of 6 or more
* Ability to supply own transportation to care receiver's home; active drivers license and automobile insurance (or alternate transportation such as city bus)

Exclusion Criteria:

* Current problem drinking
* Psychosis
* Significant cognitive impairment (MOCA<22)
* Hearing problems that preclude engagement with a care receiver
* Illiteracy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Van Orden, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic and behavioral data from interviews with the subjects. The final dataset will be stripped of identifiers prior to release for sharing; however, we will make the data and associated documentation available to users only under a data-sharing agreement as suggested by the NIH that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data from this research will be made available to the public in the University of Rochester's institutional repository, UR Research, at https://urresearch.rochester.edu. UR Research is fully searchable in its own right, and is also regularly indexed by Google, so that its contents are accessible from the results of Google searches.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication of primary outcomes
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement as suggested by the NIH that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
URL: https://urresearch.rochester.edu

REFERENCES:
- [Background] Van Orden KA, Conwell Y, Chapman BP, Buttaccio A, VanBergen A, Beckwith E, Santee A, Rowe J, Palumbos D, Williams G, Messing S, Sorensen S, Tu X. The helping older people engage (HOPE) study: Protocol & COVID modifications for a randomized trial. Contemp Clin Trials Commun. 2022 Nov 30;30:101040. doi: 10.1016/j.conctc.2022.101040. eCollection 2022 Dec. PMID 36479062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Volunteering | Life Review
Started | 146 | 145
Completed | 129 | 112
Not Completed | 17 | 33
Not completed — Death | 0 | 3
Not completed — Lost to Follow-up | 9 | 13
Not completed — Withdrawal by Subject | 8 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Volunteering | Life Review | Total
Number analyzed (Participants) | 146 | 145 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.78 (9.27) | 71.46 (8.96) | 72 (9.07)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 111 | 108 | 219
  Male | 34 | 36 | 70
  Transgender male-to-female | 1 | 1 | 2
  Transgender female-to-male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 144 | 141 | 285
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 135 | 130 | 265
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 146 | 145 | 291
UCLA Loneliness Scale [Mean (Standard Deviation); unit: units on a scale] — UCLA Loneliness Scale Version 3 assesses self-reported loneliness with 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. Some items must be reverse-coded so that higher total scores reflect greater loneliness (i.e., 1=4, 2=3, 3=2, 4=1). Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness).
  units on a scale | 49.06 (10.86) | 48.94 (9.57) | 49 (10.22)
Quality of Life (WHOQOL) [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life--Bref instrument (WHOQOL-Bref) is a self-report instrument with 26 items and a total score reflecting overall health-related quality of life. All items are rated on a 5-pt scale, with scores of 5 representing the best outcome. Some items are reversed scored (per the WHOQOL manual). Scores are transformed (per WHOQOL manual) such that the range for the total score is 0-100, with 100 representing the highest quality of life.
  units on a scale | 68.28 (13.79) | 69.29 (12.80) | 68.35 (13.57)
Belonging (Interpersonal Needs Questionnaire) [Mean (Standard Deviation); unit: units on a scale] — Perceptions of belonging will be measured with the 9 items in the "belonging" subscale of the Interpersonal Needs Questionnaire. Each item is rated on a 3-pt scale: 'not at all true for me' (0), 'somewhat true for me' (1), or 'very true for me' (2). Some items are reverse scored so that higher scores represent better outcomes (i.e., greater belonging). Scores represent a sum of all items and can range from 0 - 18. This scale assesses a secondary outcome--the psychological mechanism of social connection/support.
  units on a scale | 0.68 (0.45) | 0.67 (0.41) | 0.67 (0.43)
Meaning & Purpose (PROMIS) [Mean (Standard Deviation); unit: units on a scale] — The PROMIS Meaning and Purpose short form has 4 items, rated from 1 ('not at all'), 2 ('a little bit'), 3 ('somewhat'), 4 ('quite a bit'), and 5 ('very much'). Total scores are transformed using a T-score metric in which 50 is the mean of the reference population and 10 is the standard deviation (SD) of that population. For the Meaning and Purpose form, the reference group was a general (not clinical) population. Greater scores indicate a better outcome (i.e., greater meaning and purpose). This measure assesses a secondary outcome--the psychological mechanism of purpose/perceived usefulness.
  units on a scale | 45.15 (9.77) | 45.21 (10.47) | 45.18 (10.11)
Satisfaction with Social Roles & Activities (PROMIS) [Mean (Standard Deviation); unit: units on a scale] — Satisfaction with Social Roles and Activities (PROMIS) is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate better outcomes (i.e., greater satisfaction with social role and activities). This measure assesses a secondary outcome, the psychological mechanism of social engagement.
  units on a scale | 47.44 (7.63) | 46.31 (6.96) | 46.87 (7.31)
Social Isolation (PROMIS) [Mean (Standard Deviation); unit: units on a scale] — Social isolation (PROMIS) is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate worse outcomes (i.e., greater social isolation).
  units on a scale | 53.98 (6.31) | 54.53 (6.01) | 54.26 (6.16)

OUTCOME MEASURES:

1. Primary Outcome: Loneliness
Description: UCLA Loneliness Scale Version 3, which assesses self-reported loneliness. 20 items, rated as to how often the participant has felt a certain way in the prior month (e.g., "How often do you feel alone?") -- "never" (1), "rarely" (2), "sometimes" (3), or "often" (4). Higher scores indicate greater loneliness. However, some individual items must be reverse-coded so that higher total scores reflect greater loneliness (i.e., 1=4, 2=3, 3=2, 4=1). These items (e.g., "How often do you feel there are people you can turn to?") are items 1,5,6,9,10,15,16,19,20. Total scores range from 20 to 80, with higher scores representing a worse outcome (i.e., greater loneliness). Subjects completed this scale at 1 year follow-up, reflecting on the prior month.
Time Frame: Month 12
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
units on a scale | 44.36 (0.96) | 44.10 (1.00)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = .896, Mixed Models Analysis; Mean Difference (Final Values) = -.138, 95% CI 2-sided [-2.21 to 1.93], Standard Error of Mean 1.06

2. Primary Outcome: Health-related Quality of Life
Description: World Health Organization Quality of Life--Bref instrument (WHOQOL-Bref). This self-report instrument comprises 26 items. The WHOQOL-Bref produces scores for four domains (i.e., physical health, psychological functioning, social relationships, and environmental opportunities) and a total score reflecting overall health-related quality of life. Our primary outcome is the total score assessing overall quality of life. All items are rated on a 5-pt scale, with scores of 5 representing the best outcome. Some items are reversed scored (per the WHOQOL manual). Scores are transformed (per the WHOQOL manual) such that the range for the total score is 0-100, with 100 representing the highest quality of life.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
score on a scale | 91.82 (1.25) | 91.36 (1.33)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = 0.80, ANOVA; Mean Difference (Final Values) = 0.44

3. Secondary Outcome: Belonging (Mechanism)
Description: Perceptions of belonging will be measured with the 9 items in the "belonging" subscale of the Interpersonal Needs Questionnaire. Each item is rated on a 3-pt scale: 'not at all true for me' (0), 'somewhat true for me' (1), or 'very true for me' (2). Some items are reverse scored so that higher scores represent better outcomes (i.e., greater belonging). Scores represent a sum of all items and can range from 0 - 18.
Time Frame: Month 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
score on a scale | 5.62 (0.35) | 5.03 (0.36)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = 0.33, Mixed Models Analysis; Mean Difference (Final Values) = .59

4. Secondary Outcome: Meaning and Purpose (Mechanism)
Description: The PROMIS Meaning and Purpose short form was used to assess the degree to which subjects felt increased usefulness and purpose. It has 4 items, rated from 1 ('not at all'), 2 ('a little bit'), 3 ('somewhat'), 4 ('quite a bit'), and 5 ('very much'). Total scores are transformed using a T-score metric in which 50 is the mean of the reference population and 10 is the standard deviation (SD) of that population. For the Meaning and Purpose form, the reference group was a general (not clinical) population. Greater scores indicate a better outcome (i.e., greater meaning and purpose).
Time Frame: Month 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
score on a scale | 47.25 (0.89) | 47.07 (0.92)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Final Values) = .08

5. Secondary Outcome: Satisfaction With Social Roles and Activities (Mechanism)
Description: Satisfaction with Social Roles and Activities (PROMIS) was used to assess the construct of social engagement. It is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate better outcomes (i.e., greater satisfaction with social role and activities).
Time Frame: Month 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
score on a scale | 47.94 (0.66) | 47.15 (0.70)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Final Values) = .8

6. Other Pre Specified Outcome: Social Isolation
Description: Social isolation (PROMIS) is a computerized adaptive test (CAT). It produces T scores with a mean of 50 and standard deviation of 10. Greater scores indicate worse outcomes (i.e., greater social isolation).
Time Frame: Month 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Volunteering | Life Review
Number analyzed (Participants) | 129 | 112
score on a scale | 51.64 (0.59) | 51.72 (.62)
Statistical Analysis 1: Comparison: Volunteering vs Life Review; Test type: Superiority; p = 0.57, Mixed Models Analysis; Mean Difference (Final Values) = .08

ADVERSE EVENTS:
Time Frame: Subjects were assessed for adverse events at all study visits; participation was 1 year, with assessments at 3-months post-randomization, 6-months post randomization, 9 months post randomization, and 12-months post-randomization.
Arm/Group | Volunteering | Life Review
All-Cause Mortality (participants affected / at risk) | 0/146 | 3/145
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/145
Other Adverse Events (participants affected / at risk) | 0/146 | 0/145

LIMITATIONS AND CAVEATS:
Few participants (i.e., 9%) completed the minimum 'dose' of volunteering expected to confer benefit (i.e., at least 4 hours per month) and 30% did not begin any volunteer service. 'Dose' for the control condition was comparable. Given that few participants received a 'full dose' of study interventions, 'dose' analyses are planned to examine whether those who completed interventions demonstrated better outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT03343483/Prot_SAP_001.pdf
  • Informed Consent Form (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT03343483/ICF_000.pdf